CLINICAL TRIAL: NCT04379414
Title: Young, Empowered &Amp; Strong (YES): The Young Women's Breast Cancer Study 2- Focus on Newly Diagnosed/Metastatic Intervention
Brief Title: YES Study - Newly Diagnosed/Metastatic Intervention
Acronym: YES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-124
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Symptom, Behavioral
Keywords: Breast Cancer; Symptom, Behavioral
MeSH Terms: conditions — Breast Neoplasms; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Newly Diagnosed Automatic Symptom Information (Experimental): Eligible participants are consented and enrolled and randomized into 1 or 4 groups in the study. Randomization allocation not shared directly with participant.
  * Participants with early stage breast cancer will respond to baseline (at enrollment) and follow-up outcome surveys via. Participants will then create a personal YES portal account and automatically receive information on sexual health and vaginal dryness. Participants will also complete serial monitoring assessments in the portal.
  * YES portal assessments will be sent once a week for the first 12 weeks (each assessment will take approximately 10-15 minutes). After 12 weeks of weekly assessments in YES portal, the frequency of assessments will be changed to once every month.
  * Surveys will be sent once every 6 months for the first 3 years, then annually.
  * Participants will be asked to allow for medical record review, two blood samples (baseline and 3-6 months), and a sample of any tissue available to bank.
  Interventions: Behavioral: YES portal
- Newly Diagnosed Trigger Symptom Information (Experimental): Eligible participants are consented and enrolled and randomized into 1 or 4 groups in the study. Randomization allocation not shared directly with participant.
  * Participants with early stage breast cancer will respond to baseline (at enrollment) and follow-up outcome surveys via. Participants will then create a personal YES portal account and automatically receive information on sexual health and vaginal dryness. Participants will also complete serial monitoring assessments in the portal.
  * YES portal assessments will be sent once a week for the first 12 weeks (each assessment will take approximately 10-15 minutes). After 12 weeks of weekly assessments in YES portal, the frequency of assessments will be changed to once every month.
  * Surveys will be sent once every 6 months for the first 3 years, then annually.
  * Participants will be asked to allow for medical record review, two blood samples (baseline and 3-6 months), and a sample of any tissue available to bank.
  Interventions: Behavioral: YES portal
- Metastatic Automatic Symptom Information (Experimental): Eligible participants are consented and enrolled and randomized into 1 or 4 groups in the study. Randomization allocation not shared directly with participant.
  * Participants with early stage breast cancer will respond to baseline (at enrollment) and follow-up outcome surveys via. Participants will then create a personal YES portal account and automatically receive information on sexual health and vaginal dryness. Participants will also complete serial monitoring assessments in the portal.
  * YES portal assessments will be sent once a week for the first 12 weeks (each assessment will take approximately 10-15 minutes). After 12 weeks of weekly assessments in YES portal, the frequency of assessments will be changed to once every month.
  * Surveys will be sent once every 6 months for the first 3 years, then annually.
  * Participants will be asked to allow for medical record review, two blood samples (baseline and 3-6 months), and a sample of any tissue available to bank.
  Interventions: Behavioral: YES portal
- Metastatic Trigger Symptom Information (Experimental): Eligible participants are consented and enrolled and randomized into 1 or 4 groups in the study. Randomization allocation not shared directly with participant.
  * Participants with early stage breast cancer will respond to baseline (at enrollment) and follow-up outcome surveys via. Participants will then create a personal YES portal account and automatically receive information on sexual health and vaginal dryness. Participants will also complete serial monitoring assessments in the portal.
  * YES portal assessments will be sent once a week for the first 12 weeks (each assessment will take approximately 10-15 minutes). After 12 weeks of weekly assessments in YES portal, the frequency of assessments will be changed to once every month.
  * Surveys will be sent once every 6 months for the first 3 years, then annually.
  * Participants will be asked to allow for medical record review, two blood samples (baseline and 3-6 months), and a sample of any tissue available to bank.
  Interventions: Behavioral: YES portal

INTERVENTIONS:
Behavioral: YES portal — A web-based portal designed for access by smartphone, tablet, or laptop/desktop. The portal is designed to help monitor cancer related issues and to share self-management information, resources and potential research opportunities. The portal is also designed to create a community among participants through the yeschat.org discussion board.

SUMMARY:
This research study is being done to monitor common symptoms and behavior, and to provide supportive care information and peer support, as well as research opportunities for young women ages of 18-39 years old who have been diagnosed with stage 0-IV stage breast cancer using a web-based portal (YES), built for smartphones, tablets, and computers.

DETAILED DESCRIPTION:
This is a prospective, interventional cohort study with an embedded Phase II randomized controlled clinical trial with a parallel design.

* The research study procedures include screening for eligibility, consent, enrolled, randomization into 1 of 4 groups.
* The study interventions including the (web-based portal ) YES portal use including regular assessments, serial outcome surveys, medical record review, and tumor/blood collection.
* The YES portal is a web-based portal designed for access by smartphone, tablet, or laptop/desktop. The portal is designed to help monitor cancer related issues and to share self-management information and resources to those interested in particular issues or who score high enough on the symptom measures designed to assess and track noticeable symptoms (and thus might benefit from such), as well as to share potential research opportunities when available. The portal is also designed to create a community among participants through the yeschat.org discussion board
* Participants will be in this research study for up to 5 years with the option to opt out of portal assessment component follow-up after only 1 year.
* It is expected that about 400 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-3

  * Female
  * diagnosed with breast cancer between the ages of 18-39 years
  * less than 3 months post diagnosis date of new primary or local recurrence (prior history of other cancer is allowed as long as treated with curative intent and no evidence of disease from that cancer)
  * has not started treatment for breast cancer diagnosis yet
  * is planning to get care at DFCI
  * be fluent in and able to read English
  * have internet access on a regular basis at the time of consent that can support the web-based platform
* Stage IV

  * Female
  * initial diagnosis of breast cancer between the ages of 18-39 years
  * be fluent in and able to read English
  * have internet access on a regular basis at the time of consent that can support the web-based platform

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal dryness | 1 year
  One item regarding vaginal dryness on the BCPT will be used and grouped by moderate, quite a bit, extreme responses to define the vaginal dryness rate at 1 year. Based on historical data (from our ongoing Young Women's Breast Cancer Study), the 1-year vaginal dryness rate for the control group is assumed to be 27%. For the Phase II randomized controlled trial component of the study,it will have 85% power to detect a 10% difference in the primary endpoint with 367 patients, and would plan to recruit 408 to account for dropout (last row of the table).

SECONDARY OUTCOMES:
Socio-demographics | Up to 5 years
  Women will be asked about their race, education, employment and financial status using items selected from the Alliance Patient Questionnaire that is currently being piloted (Alliance A191401), adapted to include an item on employment status that has been tested previously in a breast cancer population and is going to be added to the next version of the Alliance Patient Questionnaire.
Financial burden | Up to 5 years
  Items adapted from the National Health Interview Survey29 and the Cancer Outcomes Research and Surveillance (CanCORS) Caregiver Study30 will be used to assess financial burden and to estimate out of pocket expenses attributed to their breast cancer diagnosis.
Smoking and alcohol use | Up to 5 years
  Smoking and alcohol use will be evaluated using items selected from the prior cohort study of young women with breast cancer and our prior Smoke Free Study
Physical Activity | Up to 5 years
  Physical activity will be assessed using a modified version of the Godin Leisure-Time Exercise Questionnaire (GLTEQ).This self-reported measure is used to estimate weekly frequencies of strenuous, moderate, and light activities. It has been modified to include average duration of activities. Weekly minutes of moderate and vigorous activity (MVPA) will be the main measure of physical activity; however weekly minutes of vigorous activity (MVA) and the average weekly frequency of mild, moderate and strenuous intensity exercise based on the Leisure Score Index (LSI) will also be examined to evaluate change in physical activity behaviors. The Godin measure will be administered at multiple timepoints and will be used to evaluate change in physical activity over time.
Mobility | Up to 5 years
  The EQ-5D-5L33, 34 is a summary measure of health status for use in evaluating health and healthcare and includes five functional dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) plus a visual analog scale (EQ-VAS) that asks participants to assess how good or bad their health is today on a 0 (worst health imaginable) -100 (best health imaginable) scale. The EQ-5D-5L will be used to generate and evaluate QALYs.
Self-Care | Up to 5 years
  The EQ-5D-5L33, 34 is a summary measure of health status for use in evaluating health and healthcare and includes five functional dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) plus a visual analog scale (EQ-VAS) that asks participants to assess how good or bad their health is today on a 0 (worst health imaginable) -100 (best health imaginable) scale. The EQ-5D-5L will be used to generate and evaluate QALYs. T
Usual Activities | Up to 5 years
  The EQ-5D-5L33, 34 is a summary measure of health status for use in evaluating health and healthcare and includes five functional dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) plus a visual analog scale (EQ-VAS) that asks participants to assess how good or bad their health is today on a 0 (worst health imaginable) -100 (best health imaginable) scale. The EQ-5D-5L will be used to generate and evaluate QALYs.
Pain and Discomfort | Up to 5 years
  The EQ-5D-5L33, 34 is a summary measure of health status for use in evaluating health and healthcare and includes five functional dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) plus a visual analog scale (EQ-VAS) that asks participants to assess how good or bad their health is today on a 0 (worst health imaginable) -100 (best health imaginable) scale.
Anxiety and Depression | Up to 5 years
  The Patient Health Questionnaire (PHQ-9)35, 36 will be used to evaluate for clinically significant depression.
  (see management strategy below for the suicidality question in particular). Distress and anxiety will be assessed using select items from the PRO-CTCAE as described below. We will also ask patients to indicate the face that best represents how they feel using a publicly available 5 emoji Likert scale
Overall Symptoms | Up to 5 years
  The Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a patient-centered, standardized self-report measure that enables patients to report symptoms and AEs. The PRO-CTCAE has demonstrated favorable validity, reliability, and responsiveness in a large heterogeneous United States sample of cancer patients undergoing treatment.37 40 PRO-CTCAE items that are salient to young women with breast cancer will be collected. The PRO-CTCAE items use conditional branching for AEs that contain multiple attributes. A modified 19-item version of the Breast Cancer Prevention Trial (BCPT) Symptom Checklist will evaluate common symptoms, including hot flashes, fatigue, sexual problems, and musculoskeletal complaints. The PROMIS 8-item Fatigue Scale will be used to assess fatigue. Sleep quality will be evaluated with the Insomnia Severity Index (ISI) as well as with a modified Self-Assessment of Sleep Survey (SASS).
Adherence to Hormonal or other Oral Therapy | Up to 5 years
  Measurement of adherence to oral therapy using a 10 item self-report medication adherence measure based on work from Voils et al. among women who report currently prescribed oral hormonal or other oral therapy
Adolescent and Young Adult (AYA) Concerns | Up to 5 years
  AYA concerns will be measured by 14 items from the AYA HOPE Study42 follow-up questionnaire that ask patients to rate their level of concern regarding a range of AYA survivorship-focused issues, including fertility, diet and nutrition, physical activity, weight management, survivorship care, recurrence concerns, and financial concerns, and we have added genetics and body image. 3 items have been added to the AYA Concerns that ask about the desire for additional information about select issues facing young women with breast cancer including about body image/beauty, smoking, and alcohol consumption.
Emotional Symptoms | Up to 5 years
  Anxiety and depression will be measured by the 14-item Hospital Anxiety and Depression Scale (HADS). This is a reliable and valid instrument that is well received by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ann H Partridge, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH
URL: https://www.dana-farber.org/research/innovations